CLINICAL TRIAL: NCT02231905
Title: Open Label, Exploratory Clinical Trial to Assess the Safety, Tolerability and Effectiveness of a Switching From Talipexole to Pramipexole
Brief Title: Safety, Tolerability and Efficacy of Switching From Talipexole to Pramipexole in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 248.544
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- BI-Sifrol® (Experimental): Tablets were administrated after switching from prior treatment of dopamine agonist (talipexole), treatment period consisted of an ascending period and a maintenance period, total duration was 4 to 12 weeks.
  Interventions: Drug: BI-Sifrol®

INTERVENTIONS:
Drug: BI-Sifrol®

SUMMARY:
Study to assess the safety, tolerability and effectiveness of a switching from Domin® (talipexole) tablet to BI Sifrol® (pramipexole) tablet in patients with Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease (included juvenile parkinsonism) and treated with talipexole (Domin®)
2. Patients who present stable symptoms and maintain the doses of talipexole and other concomitant therapy for Parkinson's disease at least last 4 weeks
3. Male or female patients aged 20 and over
4. In or out-patients
5. Patient's severity characterized as Stage 1 - 5 by Modified Hoehn & Yahr scale
6. Ability to provide written informed consent in accordance with the Good Clinical Practice (GCP), Good Post-marketing Surveillance Practice (GPMSP) and other relevant laws such as the Pharmaceutical Affairs Law

Exclusion Criteria:

1. History of hypersensitivity of pramipexole
2. Psychiatric symptoms such as confusion, hallucination, delusion, agitation, delirium and abnormal behavior
3. Subjective symptom derived from orthostatic hypotension
4. Hypotension (systolic blood pressure; 100 mmHg or less)
5. Complication such as clinically significant cardiac, renal and hepatic diseases
6. Patients who drive a car, operate a machine, work on heights or engage in other hazardous activities
7. Pregnant, possibly pregnant or female in lactation
8. Patients who are participating in other drug studies or who receive other investigational drugs within last 3 months before enrolled this study
9. Other than above, those who judged by the investigator or sub-investigator to be inappropriate as for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-01; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Number of patients who prematurely discontinued due to adverse event | up to 12 weeks

SECONDARY OUTCOMES:
Change of the sum of Unified Parkinson's Disease Rating Scale (UPDRS) Part II (activities of daily living) | up to 12 weeks
Change of the sum of UPDRS Part III (motor examination) | up to 12 weeks
Change of Modified Hoehn & Yahr scale | up to 12 weeks
Change of Clinical global impression (CGI) of efficacy | up to 12 weeks
Number of patients with abnormal changes in laboratory parameters | up to 12 weeks
Number of patients with clinically significant changes in vital signs | up to 12 weeks
  Blood Pressure, Pulse Rate
Number of patients with adverse events | up to 12 weeks
Number of patients with clinically significant changes in electrocardiogram (ECG) | up to 12 weeks